CLINICAL TRIAL: NCT02933840
Title: Using a Remote Patient Monitoring Alert System to Improve Care in Geriatric Orthopedic Trauma Patients
Brief Title: Using a Remote Patient Monitoring Alert System to Improve Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Target patient population reevaluated prior to enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Aalok Agarwala, Division Chief of General Surgery Anesthesia, Associate Director of Quality and Safety, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016P002227
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Fractures, Bone; Cardiovascular Abnormalities; Respiratory System Abnormalities; Hemorrhage
MeSH Terms: conditions — Fractures, Bone; Cardiovascular Abnormalities; Respiratory System Abnormalities; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AlertWatch (Experimental): Patients will receive standard monitoring and in addition the AlertWatch software will alert the intensive care physician if there is a value that meets criteria for alerting. The care team will be the orthopedic surgery team in addition to the intensive care physician being involved as a consultant if he/she receives an alert.
  Interventions: Device: AlertWatch
- No AlertWatch (No Intervention): Patients will receive standard monitoring without the AlertWatch software. The care team will be the orthopedic surgery team without the intensive care physician being involved as a consultant.

INTERVENTIONS:
Device: AlertWatch — AlertWatch holds 510(k) FDA clearance K15335. It is a software program that takes data present in the medical record, including vital signs and laboratory results, and determines whether it meets predetermined thresholds for alerting a clinician. These thresholds are intended to correlate with signs of acute clinical deterioration in the patient being monitored.
  Arms: AlertWatch

SUMMARY:
The purpose of this study is to determine the efficacy of a remote patient monitoring platform and alert system in reducing adverse events for hospitalized geriatric orthopedic trauma patients.

DETAILED DESCRIPTION:
Geriatric orthopedic trauma patients are a particularly vulnerable cohort due to their age and medical complexity. These patients are often admitted to a floor unit with high physician-to-patient and nurse-to-patient ratios, especially during hours of low staffing intensity (eg, nighttime and weekend hours). As a result, during hours of low staffing intensity the potential for acute deterioration with delayed reaction from the care team is significant. The investigators aim to test the efficacy of a remote patient monitoring platform to reduce adverse events in this population during hours of low staffing intensity. The platform is a software called AlertWatch. It takes laboratory and vital sign data that has been reported in the medical record and determines whether it meets a cut-off value that is concerning for patient deterioration. If the value meets that cut-off, it sends a page to a recipient clinician. The investigators will have a physician trained in intensive care receive these alerts and respond to them by evaluating the patient and, in a consultative capacity, assist the primary team, namely the orthopedic surgery service, in taking care of the patient.

Patients will be randomized to intervention and control arms at the outset of their hospitalization. Patients in the intervention arm will receive standard of care monitoring and the primary team responsible for the care of the patient will remain the orthopedic surgery service, however, in addition, the AlertWatch software will be implemented and the intensive care physician will be involved in the patient's care when there is an alert. Patients in the control arm will receive standard of care monitoring and the orthopedic surgery service will be the primary team responsible. The Investigators will measure whether the intervention reduces adverse events in the study population compared with control patients.

All patients will be enrolled consecutively at the time of admission to the hospital. The AlertWatch platform (510(k) FDA clearance K15335) has the ability to automatically detect whether a patient admitted to a bed on the orthopedic surgery service meets inclusion criteria. The platform will automatically randomize patients into the active arm or the control arm of the study. For patients randomized to the active arm, the platform will provide alert monitoring.

The Investigators will also be enrolling intensive care physicians to participate in this study. Physician participation is optional. In advance of the start of the study, they will be provided information regarding the study and an informed consent document.

The AlertWatch platform has the ability to send an alert when it detects abnormalities, particular trends, or combinations of abnormalities or trends. In this study, the Investigators will use specific threshold values to alert for abnormalities and concerning trends in patient data. When an alert is made, it will be sent to the in-house intensive care physician's regular pager. The page will display the data. Orthopedic interns will continue to monitor for patient data in the standard fashion.

The Investigators will institute a protocol in which an intensive care physician is receiving alerts from AlertWatch during nighttime and weekend hours. The intensivist will: 1.) view the alert, 2.) determine whether any subsequent action is warranted. Subsequent actions may include: 1.) reviewing the patient's chart 2.) visiting the patient and/or his/her nurse 3.) paging the orthopedic surgery team to discuss the patient's situation.

There is an extremely low risk that a patient's safety would be at all threatened in either arm of the study. Patients who are assigned to the intervention arm and the control arm will both receive the standard of care. Intervention arm patients will additionally have the AlertWatch software relaying alerts to designated providers. The software does not create new, previously non-existent data. It relays data that is already available and viewable by all providers in the medical record for the patient. Given the nature of the intervention in this study, the likelihood of any adverse events due to the intervention is extremely low.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Massachusetts General Hospital or Brigham and Women's Hospital
* Admitted to orthopedic trauma surgery service
* Admitted to a non-ICU bed (patients initially admitted to an ICU and then transferred to the non-ICU bed will be included)

Exclusion Criteria:

* Admitted to service other than orthopedic trauma surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mortality | One year
  Whether a patient experiences death during their hospitalization.
Transfer to the ICU | One year
  Whether the patient is transferred from a floor unit to the intensive care unit during their hospitalization.
Cardiac arrest | One year
  Whether the patient experiences a cardiac arrest during their hospitalization.
Rapid response team called | One year
  Whether the a rapid response team is called to assess the patient during their hospitalization.

SECONDARY OUTCOMES:
Time to ordering of blood | One year
  Time from hemoglobin < 7 to when blood product is ordered for patient during their hospitalization.
Time to ordering of fluids or vasopressors | One year
  Time from systolic blood pressure<80, diastolic<40 to when fluids or vasopressors are ordered for patient during their hospitalization.
Time to ordering of diuretics, NIPPV, or intubation | One year
  Time from oxygen saturation<90% to when diuretics, NIPPV, or intubation are ordered for patient during their hospitalization.
Time to ordering of nodal blocking agent | One year
  Time from heart rate >130 to when a nodal blocking agent (beta blocker, calcium channel blocker, digoxin, or amiodarone) is ordered for patient during their hospitalization.
Time to ordering of insulin | One year
  Time from glucose >350 or <60 to when insulin is ordered for patient during their hospitalization.
Time to ordering of diuretics or insulin/D50 | One year
  Time from potassium>6 to when diuretics or insulin/D50 is ordered for patient during their hospitalization.
Time to ordering of appropriate fluids | One year
  Time from sodium>145 or sodium<130 to when appropriate fluids are ordered for patient during their hospitalization.
Time to ordering to discontinue foley catheter | One year
  Time from foley catheter insertion to foley catheter discontinuation during their hospitalization.
Time to improvement of hemoglobin | One year
  Time from hemoglobin <7 to hemoglobin>7
Time to improvement of blood pressure | One year
  Time from systolic blood pressure<80, diastolic<40 to systolic blood pressure>80, diastolic>40
Time to improvement of oxygen saturation | One year
  Time from oxygen saturation to <90% to oxygen saturation >90%
Time to improvement of heart rate | One year
  Time from heart rate >130 to heart rate <130
Time to improvement of glucose | One year
  Time from glucose >350 or <60 to glucose <350, >60
Time to improvement of potassium | One year
  Time from potassium >6 to potassium to <6
Time to improvement of sodium | One year
  Time from sodium >145 or <130 to sodium <145, >130

CONTACTS AND LOCATIONS:
Overall Officials: Aalok V Agarwala, MD, MBA, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No